CLINICAL TRIAL: NCT06398262
Title: MA_MCS_Alar SpO2 Sensor Pilot study_2020_11181
Brief Title: Alar SpO2 Sensor Study
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Alar SpO2 sensor Pilot study
Record Dates: First submitted 2024-03-06; First posted 2024-05-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: SpO2; Nasal Alar Collapse, Bilateral; Oxygen; Measurement
MeSH Terms: conditions — Nasal Alar Collapse, Bilateral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: This study will be conducted in surgical patients in the peri-operative unit of Karolinska University Hospital (Huddinge site), Stockholm, Sweden and will focus on patients after upper abdominal surgery. In order to ensure a balanced distribution of men and women, at a minimum 40% of the total subject population will be male and 40% will be female.

SUMMARY:
BACKGROUND: As the normal functioning of the body is dependent on oxygen, low blood oxygenation is a acute problem that needs immediate attention. Measurement of blood oxygenation is therefore central to monitor patients and is usually done using light technology with a clip on the finger. Philips manufactures a measuring clip that is designed to measure oxygenation in the nasal wing instead of the finger. The advantage of this is that the nose is not affected as much as the fingers by poor blood flow in the skin, for example caused by cold. The nose is also closer to the heart and lungs than the hand, so changes in oxygenation may be detected earlier. This newer meter is an approved CE-marked product that is available for clinical use, but the next step is to investigate it systematically during and after surgery.

DETAILED DESCRIPTION:
METHODS: The study intends to include patients undergoing planned major surgery at the surgery department at Karolinska University Hospital Huddinge. Before surgery, patients will be asked and written informed consent for participation will be obtained. Within the framework of the study, measurement with the newer measurement method on the nose is planned to be done at the same time as standard measurement on the finger is performed. The research study and oxygen saturation measurement with the nasal clamp starts when the patient enters the operating room and continues until he or she leaving the post-operative ward the day after surgery, or at the latest 24 hours after the start of the operation. Apart from the use of two body oxygenation monitors, there is no impact on the treatment and care are not affected at all. Decisions and actions based on possible changes in oxygenation will be based primarily on the traditional measurement point in the finger. After completion of the study, all anesthesia nurses and all nurses from the surgical and postoperative department in Huddinge who have worked with the Alar SpO2 (saturation) sensor during the study will be invited to participate in a semi-structured interview. All nurses who express interest in participating will receive an information sheet and consent will be signed personally with the signed personally with the interviewer before the interview starts. The investigators will collect data on staff opinions regarding the use of the Alar SpO2 sensor (such as: the differences between the Alar SpO2 sensor and the finger SpO2 sensor, the advantages and disadvantages of the Alar SpO2 sensor, advantages of using dual oximetry, and potential expansion of the work with the Alar SpO2 sensor).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Standard of care for planned abdominal surgery foresees continuous SpO2 monitoring intra- and post-operatively
* Standard of care for planned abdominal surgery foresees arterial catheterization in order to aspirate blood for blood gas analysis
* Expected overnight stay in the peri-operative unit
* Able to speak and understand Swedish
* Willing and able to provide written informed consent

Exclusion Criteria:

* Body weight below 50 kg
* Procedures and/or conditions affecting the face or hands that might prevent placement of sensors
* Injury/wounds or physical malformation of sensor application sites (i.e. nose, fingers)
* Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors (self-reported)
* Nail fungus on application site
* Refusal to remove artificial nails or nail polish
* Severe dermatitis or hyperkeratosis (e.g. ichthyosis) at sensor application site
* Raynaud's disease
* Hemoglobinopathy
* Expected post operative ward stay ≤12 hrs
* Dye injections within 48 hours
* Pregnant or lactating during the study period
* Nasal intubation
* Patient is participating in another medical device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in surgical patients in the peri-operative unit of Karolinska University Hospital (Huddinge site), Stockholm, Sweden and will focus on patients after upper abdominal surgery.
  In order to ensure a balanced distribution of men and women, at a minimum 40% of the total subject population will be male and 40% will be female.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Percentage of monitoring time with a perfusion indicator >0.3% for each of the two SpO2 sensors sufficient to reliably detect desaturations of both SpO2 sensors | Through study completion, estimated within 6 months
  Percentage of monitoring time with a perfusion indicator >0.3% for each
Paired sensitivity | Through study completion, estimated within 6 months
  sensitivity of the Alar SpO2 sensor vs. sensitivity of the finger SpO2 sensor
Average time difference in desaturation detection between the Alar SpO2 sensor and the finger SpO2 sensor | Through study completion, estimated within 6 months
  calculated from desaturation onset and nadir

SECONDARY OUTCOMES:
Performance of both SpO2 sensors in comparison to a CO-oximetry | Through study completion, estimated within 6 months
  Performance will be measured bu calculating Bias, Precision, Accuracy, root mean square error (ARMS), Intra-/inter-subject variability and Limits of agreement
Detection of desaturation events | Through study completion, estimated within 6 months
  Percentage of desaturation events detected by both SpO2 sensors
Number of technical alarms for both SpO2 sensors. | Through study completion, estimated within 6 months
  Number of technical alarms for both SpO2 sensors.
Staff experience and satisfaction | Through study completion, estimated within 6 months
  System Usability Scale (SUS). The system usability scale (SUS) is a simple, ten-item attitude Likert scale giving a global view of subjective assessments of usability. Participants can score every item from 1 (strongly disagree) to 5 (strongly agree). The higher they score, the more they like the system/device.
Staff experience and satisfaction | Through study completion, estimated within 6 months
  score for the Alar SpO2 sensorQualitative evaluation of nurse experience via semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Dumitrescu, Prof. Dr., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No